CLINICAL TRIAL: NCT05192174
Title: An Open-Label Non-Randomized Phase 1 Dose Escalation and Dose Expansion Study of NIB101 in Participants With Advanced Solid Tumors
Brief Title: Study of NIB101 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: due to the reconsideration of development strategy
Sponsor: Noile-Immune Biotech, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIB101-01
Record Dates: First submitted 2021-12-24; First posted 2022-01-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NIB101 Dose Level 1 (Experimental): 1 x 10^7 cells/body as chimeric antigen receptor (CAR) positive viable cells will be administered intravenously on Day 0.
  Interventions: Biological: NIB101
- NIB101 Dose Level 2 (Experimental): 1 x 10^8 cells/body as CAR positive viable cells will be administered intravenously on Day 0.
  Interventions: Biological: NIB101
- NIB101 Expansion Cohort (Experimental): Recommended dose determined on dose escalation phase will be administered intravenously on Day 0.
  Interventions: Biological: NIB101

INTERVENTIONS:
Biological: NIB101 — NIB101

SUMMARY:
NIB101-01 study is an open-label, non-randomized Phase 1 study in participants with GM2 positive advanced solid tumor, who failed to available standard of cares to evaluate the safety and tolerability of NIB101.

DETAILED DESCRIPTION:
The screening begins by signing the informed consent form and determining the participant's initial eligibility. Alternatively, in advance, the prescreening enables participants to confirm GM2 expression using the archived samples by signing the prescreening ICF prior to the screening. After the consent is obtained and the eligibility of participants is confirmed, the participant will undergo apheresis. Lymphodepleting chemotherapy will be administered prior to NIB101 infusion. After manufacturing of NIB101, participants will receive a single dose of NIB101 intravenously on Day 0 and be followed for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant with histologically or cytologically confirmed solid tumor.
2. Participant who failed or are intolerable to available standard of cares (regardless of the number of prior lines of therapy) at the investigator's discretion.
3. Participant whose tumor tissues express GM2 membrane as determined by immunohistochemistry.
4. Participant who has measurable lesions.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Life expectancy >=12 weeks from the signing screening ICF.
7. Participant with adequate organ functions.
8. Participant who can undergo apheresis at the investigator's discretion.
9. Participant must agree to use adequate contraception methods
10. Participant who is willing to sign a written informed consent.

Exclusion Criteria:

1. Active brain metastasis on the screening MRI (in case of MRI contradiction, CT is acceptable)
2. Participant with an active, known or suspected autoimmune disease requiring immune suppressive agents other than hormonal replacement therapy.
3. Prior malignancy (other than targeted GM2 positive malignancy) within the previous 3 years the signing screening ICF.
4. Suspected malignant lymphoma or leukemia
5. Participant with known or suspected interstitial pneumonia
6. Active infections requiring treatments
7. Participant with an active, known or suspected gangliosidosis.
8. Other concurrent serious diseases that may interfere with planned study intervention per investigator's discretion.
9. Prior treatment with engineered T-cell therapy/gene therapy.
10. Prior treatment with any GM2, Interleukin-7 (IL-7) or Chemokine (C-C motif) ligand 19 (CCL19) targeted therapy.
11. Participant with a condition requiring systemic treatment with either corticosteroids (>= 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to apheresis. Inhaled or topical steroids, and adrenal replacement steroid doses <10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
12. Participant with adverse events due to prior therapy have not recovered to grade 1 or baseline, except for non-clinically significant adverse events at the investigator's discretion such as alopecia.
13. Anti-neoplasm treatment within 14 days prior to apheresis
14. Radiation therapy within 14 days prior to apheresis
15. Participant currently requiring ganciclovir, valganciclovir, and so on (the drug that provides HSV-TK substrate) treatment. Participants currently receiving prophylaxis treatment can be enrolled if the prophylaxis treatment is completed before apheresis.
16. Major surgery within 4 weeks prior to screening informed consent.
17. Prior treatment with any investigational study drug/investigational study cell and gene therapies within 28 days before signing screening ICF.
18. Positive human immunodeficiency virus (HIV) and/or Human T-cell leukemia virus-1 (HTLV-1) antibody test on the screening prior to apheresis.
19. Positive Hepatitis B surface (HBs) antigen or Hepatitis C virus (HCV) antibody test on the screening prior to apheresis. Participant who has positive HBs antibody or Hepatitis B core (HBc) antibody can be enrolled if Hepatitis B virus (HBV)-DNA is undetectable.
20. Any symptoms of suspected syphilis
21. Pregnant or breastfeeding
22. History of allergy or hypersensitivity to components of NIB101 or materials used for manufacturing NIB101.
23. Hypersensitivity or contraindicated to study intervention components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | 28 days after NIB101 infusion
  Specific adverse events defined in the protocol and related to NIB101 infusion
Adverse Events | 2 years from NIB101 infusion
  Number of participants with adverse events

SECONDARY OUTCOMES:
Objective Response | 2 years from NIB101 infusion
  Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD) determined by the investigator per RECIST version 1.1 or modified RECIST
Overall Response Rate | 2 years from NIB101 infusion
  Percentage of subjects who achieved PR or better
Disease Control Rate | 2 years from NIB101 infusion
  Percentage of subjects who achieved SD or better
Duration of Response | 2 years from NIB101 infusion
  Time from first documentation of response (PR or better) to first documentation of disease progression or death from any cause
Time To Response | 2 years from NIB101 infusion
  Time from NIB101 infusion to the initial documented response (PR or better)
Progression Free Survival | 2 years from NIB101 infusion
  Time from NIB101 infusion to the date of disease progression or death from any cause.
Overall Survival | 2 years from NIB101 infusion
  Time from NIB101 infusion to time of death due to any cause
Pharmacokinetics (Cmax) | 2 years from NIB101 infusion
  Maximum peak of NIB101
Pharmacokinetics (Tmax) | 2 years from NIB101 infusion
  Time to maximum peak of NIB101
Pharmacokinetics (T1/2) | 2 years from NIB101 infusion
  Half life of NIB101
Pharmacokinetics (Clast) | 2 years from NIB101 infusion
  Concentration of last quantified NIB101
Pharmacokinetics (Tlast) | 2 years from NIB101 infusion
  Time of Clast observed
Pharmacokinetics (AUC) | 2 years from NIB101 infusion
  Area under the curve of NIB101
Immunogenicity | 2 years from NIB101 infusion
  Evaluation of an anti-CAR antibody response
Replication Competent Retrovirus (RCR) | 2 years from NIB101 infusion
  Number of cases of positive RCR

CONTACTS AND LOCATIONS:
Overall Officials: Noile-Immune Biotech, Inc., Study Director — Noile-Immune Biotech, Inc
Locations (2):
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No